CLINICAL TRIAL: NCT06079346
Title: A Randomized Phase 2b/Phase 3 Study of the TGF-β2 Targeting Antisense Oligonucleotide OT-101 in Combination With mFOLFIRINOX Compared With mFOLFIRINOX Alone in Patients With Advanced and Unresectable or Metastatic Pancreatic Cancer
Brief Title: A Study of OT-101 With mFOLFIRINOX in Patients With Advanced and Unresectable or Metastatic Pancreatic Cancer
Acronym: STOP-PC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oncotelic Inc. (Industry)
Responsible Party: Sponsor
Organization: Mateon Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OT-01-P201
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OT-101 + mFOLFIRINOX (Active Comparator): OT-101 IV dosed on Days 4-7 plus mFOLFIRINOX (dl-LV 400 mg/m2, irinotecan 180 mg/m2 and oxaliplatin 85 mg/m2 followed by a 46-hour infusion of 5-FU 2400 mg/m2) initiated on Day 1 of a 14-day cycle
  Interventions: Drug: OT-101; Drug: mFOLFIRINOX
- mFOLFIRINOX Only (Placebo Comparator): mFOLFIRINOX (dl-LV 400 mg/m2, irinotecan 180 mg/m2 and oxaliplatin 85 mg/m2 followed by a 46-hour infusion of 5-FU 2400 mg/m2) initiated on Day 1 of a 14-day cycle
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: OT-101 — OT-101: antisense oligodeoxynucleotide complementary to the messenger ribonucleic acid (mRNA) of the human TGF-β2 gene
  Arms: OT-101 + mFOLFIRINOX
Drug: mFOLFIRINOX — Folinic acid, 5-FU, Irinotecan, Oxaliplatin

SUMMARY:
The goal of this clinical study is to compare the efficacy and safety of OT-101 in combination with mFOLFIRINOX (folinic acid, 5-FU, irinotecan, oxaliplatin) to mFOLFIRINOX alone in patients with advanced and unresectable or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OT-01-P201 is designed as a randomized, open-label, active controlled, multicenter Phase 2B/Phase 3 study designed to compare the efficacy and safety of OT-101 in combination with modified FOLFIRINOX (folinic acid, 5-FU, irinotecan, oxaliplatin) to modified FOLFIRINOX alone in patients with advanced and unresectable or metastatic pancreatic cancer. The primary endpoint of the study is overall survival and key secondary endpoints are progression-free survival and objective response rate.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of advanced and unresectable or metastatic pancreatic adenocarcinoma confirmed by:

   1. Histopathology from primary tumor in pancreas, OR
   2. Histopathology from a non-pancreatic lesion in the presence of a mass in the pancreas consistent with pancreatic adenocarcinoma or a medically documented history of pancreatic adenocarcinoma.
2. Measurable disease per RECIST v.1.1
3. Male or non-pregnant, non-lactating female, ≥18 years or age

   1. If a female patient is of child-bearing potential, as evidenced by menstrual periods, she must have a negative serum pregnancy test (beta-human chorionic gonadotropin [β- hCG]) documented prior to the first administration of stud drugs
   2. Female patients of childbearing age and women < 12 months since the onset of menopause must agree to use acceptable contraceptive methods for the duration of the study and 9 months following the last injection of OT-101.
   3. Male patients must use effective contraception for a duration of 6 months after the final dose, as per the prescribing information for oxaliplatin.
4. Provide signed written informed consent
5. Eastern Cooperative Group (ECOG) Performance Status (PS) score of 0-1
6. Willingness and ability to comply with study requirements
7. Patient has adequate organ function by the following laboratory assessments at baseline(obtained ≤28 days prior to Randomization):

   Hematologic
   * Platelets ≥100×109/L
   * Hemoglobin ≥9.0 g/dL
   * Absolute Neutrophil Count (ANC) ≥1.5×109/L
   * Patient has acceptable coagulation values obtained ≤28 days prior to Randomization as demonstrated by prothrombin time (PT) or international normalized ratio (INR) and partial thromboplastin time (PTT) ≤1.5× upper limit of normal (ULN) (if on Coumadin, patient must be changed to LMWH or on Factor II or Xa anticoagulant with a t½ of less than 24 hours

   Hepatic
   * Aspartate transaminase (AST)/alanine transaminase (ALT) ≤3×ULN (if liver metastases are present, ≤5×ULN)
   * Alkaline phosphatase ≤2.0×ULN (if liver metastases are present, ≤5×ULN)
   * Total bilirubin ≤2.0×ULN (in patients with Gilbert's Syndrome total bilirubin < or = 2.5xULN)

   Renal
   * Calculated creatinine clearance ≥50 mL/min. Actual body weight should be used for calculating creatinine clearance (e.g., using the Modification of Diet in Renal Disease [MDRD] formula. For patients with a body mass index (BMI) >30 kg/m2, lean body weight should be used instead
8. Patient must have a life expectancy of ≥3 months in the opinion of the Investigator

Exclusion Criteria:

1. Diagnosis of pancreatic islet neoplasm, acinar cell carcinoma, non-adenocarcinoma (ie,lymphoma, sarcoma), adenocarcinoma originating from the biliary tree, or cystadenocarcinoma
2. Patient has experienced a decrease in ECOG PS between Screening visit and within 72 hours prior to Randomization
3. Patient on Coumadin and not willing to change to LMWH or oral Factor II or Xa inhibitor with t½ of less than 24 hours
4. History of prior malignancy, except for adequately treated in situ cancer, basal cell, squamous cell skin cancer, or other cancers (eg, breast and prostate) for which the patient has been disease-free for at least 3 years. Patients with prior cancer that is adequately controlled per the judgement of the Investigator will not be excluded from the study
5. Any serious medical condition, laboratory abnormality, psychiatric illness, or comorbidity that, in the judgment of the Investigator, would make the patient inappropriate for the study
6. Patients with abnormal electrocardiogram (ECG) at baseline (QT or QTc interval >470 ms) will be excluded from this study. The eligibility of patients with ventricular pacemakers for whom the QT interval may not be accurately measurable will be determined on a case-by-case basis by the Sponsor's medical representative in consultation with the principal investigator.
7. Serious systemic fungal, bacterial, viral, or other infection that is not controlled or requires intravenous antibiotics
8. Known history of positivity (regardless of immune status) for human immunodeficiency virus(HIV)
9. Known history of chronic active or active viral hepatitis A, B, or C infection
10. Clinically significant bleeding within 2 weeks prior to Randomization (eg, gastrointestinal[GI] bleeding or intracranial hemorrhage)
11. Pregnant or lactating women
12. Myocardial infarction, coronary bypass surgery, or arterial thromboembolic events within the last 6 months prior to Randomization, symptomatic congestive heart failure (New York Heart Association Classification >Class II, unstable angina, or unstable cardiac arrhythmia requiring medication
13. Clinically significant ascites defined as requiring ≥1 paracentesis every 2 weeks
14. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (ie, larger than what is required for placement of central venous access, percutaneous feeding tube, or biopsy) within 28 days prior to Randomization or anticipated surgery during the study period
15. Prior history of receiving immune checkpoint inhibitors (anti-CTLA4, anti-PD1, anti-PD-L1)
16. Peripheral neuropathy (>Grade 1)
17. Known history of dihydropyrimidine dehydrogenase deficiency (DPD) - Dihydropyrimidine dehydrogenase (DPD) is the initial and rate-limiting enzyme in the catabolism of 5-fluorouracil (5-FU). Thus, patients with a DPD deficiency are at risk of developing severe 5-FU-associated toxicity
18. History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegner´s granulomatosis, Sjogren´s syndrome, Bell´s palsy, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, except for psoriasis not requiring systemic therapy, vitiligo or alopecia areata, or hypothyroidism
19. Patients receiving any of the following medications are not eligible for study:

    1. Investigational agents other than the protocol drugs
    2. Anti-coagulants (except for heparin to maintain the patency of central venous catheters)
    3. Non-steroidal anti-inflammatory drugs
    4. Clopidogrel (Plavix), dipyridamole (Persantine), or any other drug that inhibits platelet functions
    5. Patients on greater than 2 mg dexamethasone, 10 mg Prednisone or or equivalent dose in alternate corticosteroid daily or actively undergoing corticosteroid dose escalation are NOT eligible
20. History of allergic reactions or known hypersensitivity to compounds of similar chemical or biologic composition to OT-101 such as anti-sense oligonucleotides or siRNA
21. Patients who are unable to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy. Telemedicine visits are acceptable
22. Not willing and able to comply with study requirements including protocol mandated procedures and visits
23. Other contraindications as defined in the product label of the components of the mFOLFIRINOX treatment regimen
24. Participation in another investigational clinical trial within 30 days of receiving the last dose of investigational study drug
25. Clinically significant psychiatric disorders, legal incapacity or limited legal capacity
26. Patients with a primary immunodeficiency
27. Patients with active central nervous system (CNS) metastases. (Patients with adequately treated CNS metastases who are clinically stable for at least 6 weeks after discontinuation of corticosteroids may be eligible for enrollment with the approval of the Sponsor's medical representative and the principal investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 2.5 years
  To compare the efficacy of OT-101 in combination with mFOLFIRINOX versus mFOLFIRINOX alone in patients with advanced and unresectable or metastatic pancreatic cancer as measured by overall survival (OS)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter - Area Under the Curve (AUC) | 1 year
  To characterize the area under the curve (AUC) of OT-101 when it is combined with mFOLFIRINOX in patients with advanced and unresectable or metastatic pancreatic cancer. Area under the curve is a measure of how much a drug reaches a person's bloodstream in a given period of time after a dose is given.
Pharmacokinetic (PK) Parameter - Cmax | 1 year
  To characterize the Cmax of OT-101 when it is combined with mFOLFIRINOX in patients with advanced and unresectable or metastatic pancreatic cancer. Cmax is the highest concentration of a drug in the blood, cerebrospinal fluid, or target organ after a dose is given.
Progression-Free Survival (PFS) | 2.5 years
  To assess the efficacy of OT-101 in combination with mFOLFIRINOX in patients with advanced and unresectable or metastatic pancreatic cancer as measured by Progression-free survival (PFS)
Objective Response Rate (ORR) | 2.5 years
  To assess the efficacy of OT-101 in combination with mFOLFIRINOX in patients with advanced and unresectable or metastatic pancreatic cancer as measured by Objective Response Rate (ORR)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2.5 years
  To compare the incidence of treatment-emergent adverse events of OT-101 in combination with mFOLFIRINOX versus mFOLFIRINOX alone

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Karmanos Cancer Center, Detroit, Michigan
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No